CLINICAL TRIAL: NCT03863418
Title: The Use of Probiotic Lactobacillus Rhamnosus GG for Treatment of Atopic Dermatitis in Children
Brief Title: Probiotic Lactobacillus Rhamnosus GG for Pediatric Atopic Dermatitis
Acronym: PROPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 400/19
Record Dates: First submitted 2019-03-03; First posted 2019-03-05 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus rhamnosus GG (Experimental): Lactobacillus rhamnosus GG (10 billion Colony Forming Units/CAPSULE)
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG
- placebo (Placebo Comparator): maltodextrin
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — PROBIOTIC
  Arms: Lactobacillus rhamnosus GG
Other: placebo — placebo
  Arms: placebo

SUMMARY:
Atopic dermatitis (AD) is a multifactorial, chronic inflammatory skin disorder that results in areas of dry, itchy skin. AD affects up to 20% of children in Western societies and represents a prevalent, burdensome, and psychologically important pediatric concern.

It often appears in infancy and may persist into adolescence and adulthood. This complex disease is typified by defective skin barrier function with activation of abnormal immunological and inflammatory pathways upon exposure to ubiquitous environmental allergens.

It often appears in infancy and may persist into adolescence and adulthood. This complex disease is typified by defective skin barrier function with activation of abnormal immunological and inflammatory pathways upon exposure to ubiquitous environmental allergens.

This complex disease is typified by defective skin barrier function with activation of abnormal immunological and inflammatory pathways upon exposure to ubiquitous environmental allergens. This phenomenon may be primarily related to mutations in important barrier proteins, in the same fashion as filaggrin in the atopic skin, or may be secondary, reflecting the intestinal mucosal damage caused by local hypersensitivity reactions to food antigens or to microbial components as in inflammatory bowel disease. Conventional therapy for AD consists of elimination of exacerbating factors, moisturizers to maintain skin hydration, antihistamines to alleviate pruritus, topically applied corticosteroids, or topical calcineurin inhibitors to control inflammation. Severe forms of atopic dermatitis may need systemic corticosteroids, oral cyclosporine, and/or phototherapy.

Probiotics have been suggested as a novel treatment approach for atopic dermatitis. Specific probiotics have been shown to normalize intestinal permeability, to counteract intestinal immune dysfunction and to normalize gut dysbiosis. Hence, their clinical benefit may reside in the control of gut inflammation induced by various intraluminal antigens and enhancement of adaptive and especially innate immune responses.

Indeed, above and beyond balancing the gut microecology and promoting host immune defences, specific probiotics might further aid in controlling the microbial colonization of the skin, thereby reducing proneness to secondary infections which typically cause sustained symptoms. However, there are conflicting evidence on the utility of selected probiotic strains for atopic dermatitis, and major problems are due to dose and viability of strain used, duration of treatment, study population.

The aim of this randomized, double-blind, placebo-controlled study is to evaluate the efficacy of the most studied probiotic in the pediatric allergy field - Lactobacillus rhamnosus GG (LGG) - in children affected by atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-36 months
* diagnosis of Atopic Dermatitis according to SCORAD index

Exclusion Criteria

* Age < 6 months
* age > 36 months,
* skin infections,
* ichthyosis,
* food allergies,
* other allergic diseases,
* chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal and/or respiratory tract,
* administration of prebiotics/ probiotics/symbiotic/systemic immunomodulators during the 4 weeks before enrolment,
* treatments with topical immunomodulators (Tacrolimus or Pimecrolimus) over the three months prior to enrolment;
* use of corticosteroids or calcineurin antagonists or phototherapy in the previous 4 weeks,
* use of systemic antibiotics or anti-mycotic drugs during 4 weeks before study entry;
* investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements;
* participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study;
* hypersensitivity to components contained in study product.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of SCORing Atopic Dermatitis (SCORAD) | after 12-week treatment
  The efficacy of LGG supplementation on clinical course of children in terms of reduction of SCORAD index (score minimum 0 - maximum 60)

SECONDARY OUTCOMES:
Composition of gut microbiota | after 12-week treatment
  gut microbiota metagenomic in term of total genomic DNA
Composition of gut microbiota metabolomic feature | after 12-week treatment
  Determination of short chain fatty acids
evaluation acquired immunity | after 12-week treatment
  evaluation acquired immunity by determining fecal Immunoglobulin A levels
evaluation of quality of life | after 12-week treatment
  evaluation of Infant Dermatitis Quality of Life Questionnaire (IDQOL) (score minimum 0 - maximum 30)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carucci L, Nocerino R, Paparo L, De Filippis F, Coppola S, Giglio V, Cozzolino T, Valentino V, Sequino G, Bedogni G, Russo R, Ercolini D, Berni Canani R. Therapeutic effects elicited by the probiotic Lacticaseibacillus rhamnosus GG in children with atopic dermatitis. The results of the ProPAD trial. Pediatr Allergy Immunol. 2022 Aug;33(8):e13836. doi: 10.1111/pai.13836. PMID 36003050